CLINICAL TRIAL: NCT05253144
Title: Rational-MCC: A Randomised Phase III Multi-centre Trial Comparing Radical Surgery and Radical Radiotherapy as First Definitive Treatment for Primary MCC
Brief Title: Comparing Radical Surgery and Radical Radiotherapy as First Definitive Treatment for Primary MCC
Acronym: Rational-MCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Efficacy and Mechanism Evaluation (EME) Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-019
Record Dates: First submitted 2021-11-02; First posted 2022-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Phase III
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Prioritise Radiotherapy (Experimental): Radical radiotherapy to macroscopic tumour and/or to the tumour bed if already excised, plus a wide margin.
  Interventions: Radiation: Radiotherapy
- Arm B: Prioritise Surgery (Experimental): Wide Local Excision (WLE), aiming for complete excision of all MCC, plus a wide margin
  Interventions: Procedure: Surgery

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy
  Arms: Arm A: Prioritise Radiotherapy
Procedure: Surgery — Surgery
  Arms: Arm B: Prioritise Surgery

SUMMARY:
A randomised phase III multi-centre trial comparing radical surgery and radical radiotherapy as first definitive treatment for primary MCC

DETAILED DESCRIPTION:
A randomised phase III multi-centre trial comparing radical surgery and radical radiotherapy as first definitive treatment for primary MCC with an observational study for patients ineligible for the randomised trial.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria for All Patients:

1. Patients newly diagnosed with histologically-proven MCC (either primary and/or regional nodal disease)
2. Completion of clinical and radiological staging investigations, including CT imaging (or other modality) of regional nodal basin(s) and major viscera (and SLNB if clinically appropriate) to identify regional and distant metastases
3. No confirmed distant metastases beyond the regional nodal basin (i.e. not stage IV disease)
4. Suitable for radical treatment to achieve disease control
5. Able to give valid informed consent
6. Consent for collection of data and tissue samples and follow up
7. Life expectancy six months or greater in relation to general fitness and co-morbidities

Additional Inclusion Criteria for Rational Compare:

1. Patients newly diagnosed with histologically-proven primary MCC
2. In the opinion of the SSMDT, the primary MCC can be encompassed both within a wide surgical margin and within a radiotherapy field, and the SSMDT is in equipoise regarding WLE or radiotherapy as first treatment
3. A minimum margin of 1 cm surrounding the MCC achievable by either radiotherapy or surgery
4. Consent for randomisation into Rational Compare

Exclusion Criteria:

1. The primary MCC has already been treated radically with WLE (surgical margins >10 mm) or radiotherapy
2. Intended use of regional or systemic chemotherapy for MCC (including molecularly targeted agents and immunotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03-19 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Time to loco-regional failure | Time from randomisation to 3 years
  The time to loco regional failure for all patients is the time from randomisation to loco-regional treatment failure

SECONDARY OUTCOMES:
The proportion of patients alive and free of loco-regional disease | Time from randomisation to 3 years
  (irrespective of whether loco-regional failure has been previously demonstrated)
Time to 'local failure'-the time from randomisation to macroscopic persistence, progression or recurrence between the primary site and regional nodal basin(s) | Time from randomisation to 3 years
  (including in-field and in transit metastases)
Time to regional nodal failure | Time from randomisation to 3 years
  Time to regional nodal failure
Time to distant progression | Time from randomisation to 3 years
  Time to distant progression
Patient Progression free survival | Time from randomisation to 3 years
  Patient Progression free survival
Patient survival | Time from randomisation to 3 years
  Survival from randomisation
Quality of life assessed by questionnaires | Time from randomisation to 3 years
  Quality of life assessed by QLQC30/ EQ-5L-5D questionnaire completion

CONTACTS AND LOCATIONS:
Overall Officials: Neil Steven, Principal Investigator — University of Birmingham
Locations (14):
- United Kingdom (14):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Tayside, Dundee
  - Barts Health NHS Trust, London
  - Christie NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - St Helens and Knowsley Hospitals NHS Trust, Prescot
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital of North Midlands Trust, Stoke-on-Trent
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: No